CLINICAL TRIAL: NCT06201897
Title: Comparison of Pre- and Post- Therapy Real Time Cortical Excitability in West Syndrome Using Transcranial Magnetic Stimulation: A Longitudinal Cohort Study
Brief Title: Cortical Excitability in West Syndrome Using Transcranial Magnetic Stimulation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, PROFESSOR, All India Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IECPG156/24.03.2022-OT-12.2023
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: West Syndrome
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Other): Children receiving ACTH therapy for West Syndrome
  Interventions: Drug: ACTH/Oral Steroids

INTERVENTIONS:
Drug: ACTH/Oral Steroids — Injection ACTH or Oral Steroids in children with West Syndrome
  Other Names: Hormonal Therapy

SUMMARY:
Currently, no literature is available regarding degree of cortical excitability and its correlation with various epileptic syndromes and disorders such as West Syndrome in pediatric age group. Studying the complex interaction of cortical excitability, seizures, neurobehavioral patterns and brain maturation in children may provide valuable information and new insights about the underlying neuropathogenic pathways in childhood epilepsy. West Syndrome is a unique epilepsy syndrome amalgamating infantile onset epilepsy with significant neurodevelopmental delay. Due to this reason, it is the ideal disorder to study this complex interaction. How cortical excitability correlates with disease activity in West Syndrome is speculative. The ability of disease characteristics such as degree of cortical excitability to predict successful outcome after ACTH therapy (non-invasive biomarker of treatment response) in children with West Syndrome has not been explored.

Most importantly, the present study may be a hypothesis generating initial step bringing new insights into neurocognitive effects of seizures, seizure pathogenesis, individualized antiepileptic drug therapy and for studying treatment response.

The investigators aim to determine the change in cortical excitability pre and post ACTH therapy, in children with West syndrome and whether the change predicts responsiveness to ACTH therapy, in terms of reduction in spasm frequency at 12 weeks.

DETAILED DESCRIPTION:
PATIENT ENROLLMENT AND MANAGEMENT:

* Consecutive children with West Syndrome (clinical spasm with EEG correlate) will be screened in the study centre for eligibility, and after applying inclusion and exclusion criteria they will be worked up for etiology.
* History will be taken and clinical examination will be done and if either are suggestive of any underlying etiology specific investigations will be performed as indicated (Ex. Neurocutaneous markers in tuberous sclerosis).
* If there are no other etiological pointers available from history and examination or if there is any history suggestive of adverse perinatal events, MRI brain with epilepsy protocol will be done.
* If MRI is not suggestive of structural etiology, they will be given a vitamin trial (pyridoxine 30mg/kg/day, pyridoxal phosphate- 20mg/kg/day, biotin 10mg/day and folinic acid 15mg/day) for a period of 10 days for response. Those who respond to vitamin trial will be excluded from the study.
* Written informed consent will be taken from legal guardians who are willing to participate in the study. Their anti-epileptic drugs will be optimized. Inappropriate AEDs like phenytoin, phenobarbitone and carbamazepine will be discontinued and replaced with valproate/levetiracetam and clonazepam in adequate doses and will be made in tablet form.
* DASII will be administered by child psychologist and will be repeated at 6 months of follow-up wherever feasible.

ACTH therapy

* Appropriate screening for Tuberculosis as per unit protocol (Mantoux and CXR screening) will be done if going to receive ACTH therapy.
* Children fulfilling the inclusion and exclusion criteria, will be enrolled and started on high dose regimen of 150 U/m2 or 6 U/kg of ACTH.
* This high dose will be continued for 2 weeks following which they will be slowly tapered over remaining 4 weeks, for a total treatment duration of 6 weeks.
* RBS and BP monitoring to be done twice weekly.
* EEG and TMS parameters will be done at baseline, 6 weeks and 3 months of therapy.
* First follow-up will be at 6 weeks of treatment initiation, then at 8 weeks and from then on once a month for a minimum period of 3 months (+/- 7 days) upto 6 months (+/- 7 days) wherever feasible.
* Those who have had complete electroclinical spasm cessation will be continued of oral AEDs.
* The overall spasm reduction will be calculated from the mean number of spasms from the observation period week and the mean number of spasms from the 6th week of therapy. Adverse effects will be noted down in their seizure diary.
* For sustained electroclinical cessation those who had complete electroclinical response will be rechecked at the end of 3 months (+/- 7 days) upto 6 months (+/- 7 days) wherever feasible.
* Compliance rate, adverse events, >50% spasm reduction rate, clinical spasm cessation rate, complete electroclinical spasm cessation rate will also be calculated from patient seizure log and EEG correlate.
* After 3 months, those who have >/=50% spasm reduction rate will be given trial of other oral AEDs as per protocol.
* But those who have <50% spasm reduction rate will be given an option to choose between ketogenic diet and vigabatrin.

KD therapy

* Children who have <50% spasm reduction rate, and opt for ketogenic diet, will be explained and counselled regarding the process of initiation and maintenance of dietary therapy.
* A window period of 5 to 7 days will be given for the pre-initiation of KD workup which includes ECG, RFT, LFT, CBC, Lipid profile, Urine calcium creatinine ratio and USG KUB for nephrocalcinosis.
* Children will be admitted in ward and initiated on Ketogenic diet under supervision.
* KD will be initiated in a ratio of 2:1 and then hiked to 2.5:1 in the next day and subsequently to 3: on day 3. Urine ketones will be checked daily using ketone dipsticks.
* For better assurance of ketosis and tolerance the indigenous KD will be supplemented with readymade formula for the initial period of 4 weeks after starting KD and then shifted to complete indigenous KD gradually over 1 week.
* If ketosis is not achieved by day 5 of starting KD, the ratio will be hiked to a maximum of 4:1 from day 6.
* Patient will be discharged as soon as the desired ratio of KD is achieved, and the parents are adequately motivated and confident. Telephonic contacts will be made in regular intervals to further ensure compliance at home.
* Those children who are unable to tolerate taking adequate ketogenic diet therapy requiring discontinuation of therapy, will be considered as deviates.
* The overall spasm reduction will be calculated from the mean number of spasms from the observation period week and the mean number of spasms from the 6th week of KD therapy.
* Failure of KD: Children with response rate if not >50% spasm reduction by 6 weeks or no electroclinical cessation of spasm by 3 months, will be considered to have failed KD and shifted to standard anti-seizure medications as per protocol.
* KD will be continued if there is more than 50% spasm reduction.
* EEG and TMS will be done at 6 weeks and 3 months of KD therapy in case of clinical spasm cessation and wherever clinically indicated.
* First follow-up will be at 6 weeks of KD treatment initiation, 8 weeks and then once monthly for a minimum period of 3 months and 6 months wherever feasible. For sustained electroclinical cessation those who had complete electroclinical response will be rechecked at the end of 3 months (+/- 7 days) upto 6 months (+/- 7 days) wherever feasible.
* Compliance rate, adverse events, >50% spasm reduction rate, clinical spasm cessation rate, complete electroclinical spasm cessation rate will also be calculated from patient seizure log and EEG correlate.
* Formula based KD would be supplied to the patient free of cost. But the company will play no part in the study design, conduct, data collection or analysis.

TMS Intervention Protocol:

PARAMETERS METHODS Resting Motor Threshold (MT) - Single pulse TMS Site of stimulation - Motor Cortex Coil type- Circular coil MCF-125 (Coil outer diameter: 121 mm; Transducer head: 140.5 x 41.5 mm) Hemisphere - Bilateral hemisphere EMG recording - Contralateral APB muscle

Short interval cortical inhibition (SICI) - Paired pulse TMS in dominant hemisphere ISI - 3 msec Conditioning pulse - 80% of MT Test stimulus - 120% of MT

Long interval cortical inhibition (SICI) - Paired pulse TMS in dominant hemisphere ISI - 100 msec Conditioning pulse - 120% of MT Test stimulus - 120% of MT

Total Time Duration - 30 min The TMS will be given by machine make Magventure model no X100 with Magoption made in Denmark with standard circular coil as mentioned above.

Data Management and Analysis Data recording would be done in a Microsoft Excel spreadsheet (Microsoft Office, Microsoft Corp., Seattle, WA, USA).

Descriptive: Mean/Median/Range/Standard Deviation/Frequencies would be used to describe the demographic profile of participants and their comorbidities Comparative: A comparison between the two groups would be done. Categorical variables would be compared using Chi square/ Fischer's exact test. Depending upon the distribution of continuous variables -

* Student "t" test would be used for parametric variables.
* Mann Whitney U test would be used for nonparametric variables. Differences with p value of 0.05 or lower will be considered significant. Ethical aspects Ethical clearance: The study will be conducted after obtaining Ethical clearance from the Institute Ethical Committee.

Essentiality and Justification for the study: This study would be beneficial in generating a hypothesis as an initial step bringing new insights into seizure pathogenesis, planning individualized antiepileptic drug therapy and studying treatment response.

Consent: Patients will be enrolled only after obtaining informed written consent from the parents/guardians.

Privacy and confidentiality: Confidentiality of the records will be maintained. The parents/guardians will have full authority to enroll or withdraw the child from the study and this will not affect the future care and treatment given to the child in our hospital.

Costs of the investigations and therapy Investigations such as EEG and TMS whenever required will be done at no additional cost.

Immunotherapy which is the standard of care will be provided to the patient. All children included in the study would be examined in detail and the investigations and standard of care would be advised after they have fulfilled the inclusion criteria. Since, the investigators would be following the standard of care in every child, hence, every child enrolled would be benefitted.

The side effects and details of the investigations and intervention shall be explained to the parents in the language they understand the best and consent will be taken accordingly.

ELIGIBILITY:
Inclusion Criteria:

* • Children, aged 6 months - 2 years with electroclinical diagnosis of West syndrome

  * Sleep EEG available within last 1 week before screening.
  * Screen for tuberculosis (Chest X-ray PA view and Mantoux testing) negative
  * Parents willing for ACTH or Ketogenic Diet therapy

Exclusion Criteria:

* Already on ACTH, prednisolone vigabatrin or KD therapy > 5days
* Tuberous sclerosis
* Vitamin trial responsiveness
* Known Pre-existing contraindications for KD (IEM, Porphyria etc.)
* Chronic systemic illness (Ex: Chronic kidney disease, congenital heart diseases etc)
* Parents refusing consent for enrolment in the study.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Cortical Excitability | 12 weeks
  Change in cortical excitability in terms of Transcranial magnetic stimulation parameters like Resting Motor Threshold, Long Interval Cortical Inhibition, Short Interval Cortical Inhibition

CONTACTS AND LOCATIONS:
Overall Officials: SHEFFALI GULATI, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No